CLINICAL TRIAL: NCT01614847
Title: Tear Osmolarity Changes After Instilling Isotonic Hyaluronate Artificial Tears
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas O Salmon, OD, PhD (Other)
Responsible Party: Sponsor-Investigator, Thomas O Salmon, OD, PhD, Professor, Northeastern State University
Organization: Northeastern State University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NSUOCO-2012-11
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Results first posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Dry Eye
Keywords: dry eye; artificial tears; tear osmolarity; residence time
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Isotonic hyaluronate artificial tear (Experimental): At random, subjects will receive isotonic hyaluronate artificial tear or a control (normal saline).
  Interventions: Drug: Artificial tears
- Normal saline (Placebo Comparator)
  Interventions: Drug: Artificial tears

INTERVENTIONS:
Drug: Artificial tears — At random, subjects will receive isotonic artificial tear or a control (normal saline).

SUMMARY:
Background:

Osmolarity is defined as the concentration of particles dissolved in a solution. Normal tears contain various dissolved particles including proteins, salts and other electrolytes. The investigators plan to investigate how osmolarity of the tear film changes over time after instillation of artificial tears containing hyaluronate. This is one kind of artificial tear that is used to treat dry eye.

Dry eye and tear osmolarity:

Dry eye is a significant health problem, but diagnosis and treatment are often ambiguous and ineffective. There has been a resurgence of interest and research in dry eye in the past 5 years, and tear osmolarity has emerged as perhaps, one of the most effective ways to evaluate tear quality and dry eye status. Dry eye is usually treated with artificial tears, and many formulations are available. The investigators will test an isotonic solution that contains hyaluronate. Hyaluronate binds water and should help to maintain water on the eye.

Objective:

We plan to study the time course of possible changes in tear film osmolarity following instillation of an isotonic artificial tear containing hyaluronate. The investigators will use the TearLab, a new clinical instrument that has been developed to quickly and easily measure tear film osmolarity. Understanding how artificial tears affect tear film osmolarity over time can help doctors determine efficacy and dosing schedules. The investigators will test the isotonic hyaluronate (Blink Contacts) artificial tears relative to normal saline solution.

Hypothesis:

The investigators should be able to measure a decrease in tear osmolarity over time following instillation due to the water-binding effect of hyaluronate artificial tears relative to a control (normal saline solution).

DETAILED DESCRIPTION:
ABSTRACT:

Introduction: Tear hyper-osmolarity may be a fundamental cause of dry eye in many cases. Hyaluronate is an agent used in some artificial tears, which binds water and can protect against evaporation. It may therefore be an effective treatment for tear hyper-osmolarity.

Purpose: Our purpose was to measure changes in tear osmolarity over time following instillation of Blink Contacts, an isotonic ocular lubricant containing hyaluronate. We hypothesized that even in isotonic solution, the water-binding properties of hyaluronate would reduce tear osmolarity. This will help us better understand efficacy of this treatment and develop a rational basis for dosing schedules.

Methods: After baseline osmolarity measurements, eight subjects received either Blink Contacts or normal saline drops in both eyes. We re-measured osmolarity five minutes later, and then at 15-minute intervals up to 95 minutes. Subjects also rated comfort at each time. The next day, the experiment was repeated with the alternate drops for each subject.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age Normal vision in both eyes (20/30 best corrected) Preference for patient with dry eye symptoms

Exclusion Criteria:

* No ocular disease other than dry eye Currently taking no ocular or systemic medications that might affect results

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas O Salmon, OD, PhD, Study Director — Northeastern State University
Locations (1):
- Northeastern State University, Tahlequah, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A convenience sample of 8 subjects was recuitted from among the student population at the NSU Oklahoma College of Optometry during May-June 2012.
Pre-assignment Details: Subjects were assigned random ID numbers in preparation for assignment into the two groups. Half (4 subjects) chosen at random, would be assigned to Group 1, and receive Drop A on Day 1, then return 24 hours (Day 2) later to received Drop B. The other 4 subjects would be assigned to Group 1, and receive Drop B on Day 1 and Drop A on Day 2.
Groups:
- Group 1: Four Subjects Who Received Drop A on Day 1: All eight subject received Drop A (hyaluronate) on one day and Drop B (saline) on the other day. Subjects #1, 2, 3, 4 received Drop A on Day 1 and Drop B on Day 2.
- Group 2: Four Subjects Who Received Drop B on Day 1: All eight subject received Drop A (hyaluronate) on one day and Drop B (saline) on the other day. Subjects #5, 6, 7, 8 received Drop B on Day 1 and Drop A on Day 2.
Period: Day 1
Arm/Group | Group 1: Four Subjects Who Received Drop A on Day 1 | Group 2: Four Subjects Who Received Drop B on Day 1
Started | 4 (Four subjects chosen at random received Drop A (hyaluronate) during Day 1.) | 4 (The other 4 subjects, not to Group 1, received Drop B (saline) on Day 1.)
Completed | 4 | 4 (See Arm 1 comments.)
Not Completed | 0 | 0
Period: Day 2 (24 Hours Later)
Arm/Group | Group 1: Four Subjects Who Received Drop A on Day 1 | Group 2: Four Subjects Who Received Drop B on Day 1
Started | 4 (On Day 2, these subject will received Drop B (normal saline).) | 4 (On Day 2, these subjects received Drop A (hyaluronate).)
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1. Isotonic Hyaluronate Artificial Tear FIRST: Per sequence. Four subject, chosen at random, will receive isotonic hyaluronate artificial tear in Session 1. After a 24-hour washout period, they will return for Session 2, when they will receive saline eye drops.
- Arm 2. Normal Saline FIRST: Per sequence. The four remaining subject (see comments to left), will receive saline eye drops in Session 1. After a 24-hour washout period, they will return for Session 2, when they will receive isotonic hyaluronate artificial tears.
- Total: Total of all reporting groups
Arm/Group | Arm 1. Isotonic Hyaluronate Artificial Tear FIRST | Arm 2. Normal Saline FIRST | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.8 (1.5) | 28.0 (4.8) | 26.9 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Osmolarity Change From Baseline (mOsms/L) as a Function of Time (Minutes)
Description: Raw data: Baseline (pre-instillation) tear osmolarity was measured for right and left eyes for each subject. Then measurements were repeated at 7 times (5, 20, 35, 50, 65 890 and 95 minutes) after instillation. Data processing: 1) Baseline osmolarity was subtracted from each post-baseline measurement to give a change-from-baseline values. 2) Right and left eye change values averaged to give a mean osmolarity change for each subject at each of the seven times. 3) Mean osmolarity changes values were averaged across 8 subjects for each of the 7 times and entered in the table below. Row 1 is for Drop A (hyaluronate); Row 2 for Drop B (saline). Column are for the 7 times.
Time Frame: Baseline, followed by 7 measurements made after instillation (5, 20, 35, 50, 65, 80, 95 minutes post-instillation).
Population: Eight subjects recruited from among students at the NSU Oklahoma College of Optometry, including 6 males and 2 females who were at least 18 years of age and who had no known ocular or systemic disease other than dry eye. Six subjects did not have dry eye and 2 were diagnosed with dry eye based on Ocular Surface Disease Index (OSDI) survey scores.
Measure: Mean (Standard Error); unit: mOsmols/L
Units Other Than Participants: Eyes
Groups:
- 5 Minutes: Mean* change in tear osmolarity (mOsmol/L) from baseline 5 minutes after instillation of Drop A (Blink Contacts; hyaluronate) for each subject. (*Mean of change values measured for right and left eyes.)
- 20 Minutes: Mean* change in tear osmolarity (mOsmol/L) from baseline 20 minutes after instillation of Drop A (Blink Contacts; hyaluronate) for each subject. (*Mean of change values measured for right and left eyes.)
- 35 Minutes: Mean* change in tear osmolarity (mOsmol/L) from baseline 35 minutes after instillation of Drop A (Blink Contacts; hyaluronate) for each subject. (*Mean of change values measured for right and left eyes.)
- 50 Minutes: Mean* change in tear osmolarity (mOsmol/L) from baseline 50 minutes after instillation of Drop A (Blink Contacts; hyaluronate) for each subject. (*Mean of change values measured for right and left eyes.)
- 65 Minutes: Mean* change in tear osmolarity (mOsmol/L) from baseline 65 minutes after instillation of Drop A (Blink Contacts; hyaluronate) for each subject. (*Mean of change values measured for right and left eyes.)
- 80 Minutes: Mean* change in tear osmolarity (mOsmol/L) from baseline 80 minutes after instillation of Drop A (Blink Contacts; hyaluronate) for each subject. (*Mean of change values measured for right and left eyes.)
- 95 Minutes: Mean* change in tear osmolarity (mOsmol/L) from baseline 95 minutes after instillation of Drop A (Blink Contacts; hyaluronate) for each subject. (*Mean of change values measured for right and left eyes.)
Arm/Group | 5 Minutes | 20 Minutes | 35 Minutes | 50 Minutes | 65 Minutes | 80 Minutes | 95 Minutes
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8
Number analyzed (Eyes) | 16 | 16 | 16 | 16 | 16 | 16 | 16
mOsmols/L
  Drop A | -0.94 (0.62) | 7.25 (1.49) | 5.31 (2.19) | -4.25 (1.26) | 7.5 (1.61) | 2.31 (1.54) | 9.25 (1.39)
  Drop B | -0.8 (0.97) | -2.1 (1.43) | 2.5 (2.09) | 4.4 (1.35) | 4.9 (1.31) | 1.9 (1.32) | 8.6 (1.9)
Statistical Analysis 1: Comparison: 5 Minutes; Drop A: Mean change in osmolarity from baseline H0: No osmolarity change from baseline (e.g. mean change = 0) H1: Significant osmolarity change from baseline (mean change ≠ 0); Test type: Equivalence — Two tailed, alpha = 0.05; p = 0.4, Wilcoxon (Mann-Whitney); df=7
Statistical Analysis 2: Comparison: 20 Minutes; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — two-tailed, alpha = 0.05; p = 0.109, Wilcoxon (Mann-Whitney); df=7
Statistical Analysis 3: Comparison: 35 Minutes; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Two tailed, alpha = 0.05; p = 0.779, Wilcoxon (Mann-Whitney); df=7
Statistical Analysis 4: Comparison: 50 Minutes; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Two tailed, alpha = 0.05; p = 0.262, Wilcoxon (Mann-Whitney); df=7
Statistical Analysis 5: Comparison: 65 Minutes; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Two tailed, alpha = 0.05; p = 0.150, Wilcoxon (Mann-Whitney); df=7
Statistical Analysis 6: Comparison: 80 Minutes; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Two tailed, alpha = 0.05; p = 0.726, Wilcoxon (Mann-Whitney); df=7
Statistical Analysis 7: Comparison: 95 Minutes; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Two tailed, alpha = 0.05; p = 0.055, Wilcoxon (Mann-Whitney); df=7
Statistical Analysis 8: Comparison: 5 Minutes; Drop B: Mean change in osmolarity from baseline H0: No osmolarity change from baseline (e.g. mean change = 0) H1: Significant osmolarity change from baseline (mean change ≠ 0); Test type: Equivalence — Two tailed, alpha = 0.05; p = 0.945, Wilcoxon (Mann-Whitney); df=7
Statistical Analysis 9: Comparison: 20 Minutes; [analysis description as in outcome 1, analysis 8]; Test type: Equivalence — Alpha = 0.05; p = 0.844, Wilcoxon (Mann-Whitney); df=7
Statistical Analysis 10: Comparison: 35 Minutes; [analysis description as in outcome 1, analysis 8]; Test type: Equivalence — Two tailed, alpha = 0.05; p = 0.945, Wilcoxon (Mann-Whitney) — df=7
Statistical Analysis 11: Comparison: 50 Minutes; [analysis description as in outcome 1, analysis 8]; Test type: Equivalence — Two tailed, alpha = 0.05; p = 0.383, Wilcoxon (Mann-Whitney) — Alpha = 0.05; df=7
Statistical Analysis 12: Comparison: 65 Minutes; Mean change in osmolarity from baseline. H0: No change (e.g. mean change = 0) H1: Significant change (mean change ≠ 0); Test type: Equivalence — Two tailed, alpha = 0.05; p = 0.383, Wilcoxon (Mann-Whitney); df=7
Statistical Analysis 13: Comparison: 80 Minutes; [analysis description as in outcome 1, analysis 8]; Test type: Equivalence — Two tailed, alpha = 0.05; p = 0.672, Wilcoxon (Mann-Whitney); df=7
Statistical Analysis 14: Comparison: 95 Minutes; [analysis description as in outcome 1, analysis 8]; Test type: Equivalence — Two tailed, alpha = 0.05; p = 0.107, Wilcoxon (Mann-Whitney); df=7
Statistical Analysis 15: Comparison: 5 Minutes; Comparison of Drop A versus Drop B change in osmolarity at this point in time. H0: No difference in osmolarity change between Drop A and B (Drop A = Drop B) H1: Significant difference in osmolarity change between Drop A and Drop B; Test type: Equivalence — Two tailed, alpha = 0.05; p = 0.64, Wilcoxon (Mann-Whitney); df=12
Statistical Analysis 16: Comparison: 20 Minutes; [analysis description as in outcome 1, analysis 15]; Test type: Equivalence — Two tailed, alpha = 0.05; p = 0.040, Wilcoxon (Mann-Whitney); df=14
Statistical Analysis 17: Comparison: 35 Minutes; [analysis description as in outcome 1, analysis 15]; Test type: Equivalence — Two tailed, alpha = 0.05; p = 0.20, Wilcoxon (Mann-Whitney); df=12
Statistical Analysis 18: Comparison: 50 Minutes; [analysis description as in outcome 1, analysis 15]; Test type: Equivalence — Two tailed, alpha = 0.05; p = 0.150, Wilcoxon (Mann-Whitney); df-=12
Statistical Analysis 19: Comparison: 65 Minutes; [analysis description as in outcome 1, analysis 15]; Test type: Equivalence — Two tailed, alpha = 0.05; p = 0.730, Wilcoxon (Mann-Whitney); df=12
Statistical Analysis 20: Comparison: 80 Minutes; [analysis description as in outcome 1, analysis 15]; Test type: Equivalence — Two tailed, alpha = 0.05; p = 0.89, Wilcoxon (Mann-Whitney); df=12
Statistical Analysis 21: Comparison: 95 Minutes; [analysis description as in outcome 1, analysis 15]; Test type: Equivalence — Two tailed, alpha = 0.05; p = 0.89, Wilcoxon (Mann-Whitney); df=12

ADVERSE EVENTS:
Groups:
- Isotonic Hyaluronate Artificial Tear: At random, subjects will receive isotonic hyaluraonate artificial tear or a control (normal saline).
- Normal Saline: Subject not assigned to Arm1 (experimental group) were assigned to this group during Session 1. Twenty-four hours later subjects were assigned to the alternate groups (cross-over).
Arm/Group | Isotonic Hyaluronate Artificial Tear | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No